CLINICAL TRIAL: NCT04608175
Title: The Efficacy of Acupuncture as a Complementary Treatment for Pain and Anxiety After Breast Cancer Surgery: Pragmatic Randomized Control Trial
Brief Title: The Efficacy of Acupuncture as a Complementary Treatment for Pain and Anxiety After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Ramon Llull (Other)
Collaborators: Hospital Quiron Sagrado Corazon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001; 2019/59-FIS-HUSC (Other: Hospital Sagrado Corazón)
Record Dates: First submitted 2020-10-09; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-09

CONDITIONS: Acupuncture Therapy; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): The experimental group will receive the standard treatment administered in these cases (analgesic regimen and nursing care procedures), in addition to the following acupuncture therapy.
  In the first visit (preoperative), the anamnesis and energy diagnosis of each patient will be carried out following the practices of Traditional Chinese Medicine (TCM) to design a personalized treatment based on the patient's medical history. A treatment of approximately 10 to 12 acupuncture points will be designed considering the TCM diagnosis and medical history of each patient. Both TCM diagnosis and the points used will be reassessed in each session. The points belonging to the upper extremity of the affected breast will be treated on the contralateral side, taking care not to insert any needle in the limb on the affected side. No points in the operated region will be used.
  Interventions: Other: Acupuncture
- Control group (No Intervention): The control group will only receive standard care procedures (analgesic regimen and nursing care procedures), although they will have the same follow up visits as the patients in the intervention group to facilitate analysis of the study variables.

INTERVENTIONS:
Other: Acupuncture — Treatment of disease by inserting needles along specific pathways or meridians. The placement varies with the disease being treated. It is sometimes used in conjunction with heat, moxibustion, acupressure, or electric stimulation.
  Arms: Acupuncture group

SUMMARY:
Background: Breast cancer is one of the most prevalent cancers worldwide. Fortunately, survival has improved in recent years thanks to its early detection and curative treatments such as mastectomy. However, this medical procedure is associated with a range of unwanted effects such as postoperative pain and anxiety. Some studies have reported that acupuncture could be an effective treatment to control these types of symptoms, although only few studies have been conducted on women undergoing mastectomy.

Methods: This is a pragmatic randomized controlled trial with blind assessors. The study will be conducted in the Breast Unit of Hospital Universitario Sagrado Corazon of Barcelona (Spain). A sample of 40 women will be recruited and randomized to receive acupuncture treatment in addition to standard care procedures, or standard care procedures alone. The main outcome, pain, will be assessed after the surgical intervention and 4, 10 and 30 days later using the numerical rating scale. Secondary outcomes include anxiety, use of analgesics, nausea, adverse effects, and surgical complications.

Discussion: Acupuncture is a low-cost non-pharmacological strategy. This study will help to clarify its possible role in controlling post-mastectomy adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Primary breast cancer patient
* Candidate for breast cancer surgery (mastectomy)
* Aged between 20 and 70 years old
* Consenting to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Have a previous history of breast cancer
* Have a previous diagnosis of a severe psychiatric disorder
* Present risk factors associated with breast cancer
* Do not speak Spanish or Catalan
* Are currently participating in another trial.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Post-intervention pain at 12 hours after surgery | 12 hours after surgery (before the acupuncture treatment)
  Pain will be evaluated using the numerical rating scale (NRS). This measure uses a scale of 0 to 10 in which the higher values represent the most severe pain.
Post-intervention pain at 48 hours after surgery | 48 hours after surgery (after the acupuncture treatment)
  Pain will be evaluated using the numerical rating scale (NRS). This measure uses a scale of 0 to 10 in which the higher values represent the most severe pain.
Post-intervention pain at first out-patient visit | In the first out-patient visit between 10 and 12 days after the intervention (evaluated before the acupuncture session)
  Pain will be evaluated using the numerical rating scale (NRS). This measure uses a scale of 0 to 10 in which the higher values represent the most severe pain.
Analgesic compsumption during hospital stay | During the hospital stay
  Amount of analgesic medication administered (ex: mg)
Analgesic compsumption at home | From discharge until day 15 after surgery.
  Amount of analgesic medication administered (ex: mg)

SECONDARY OUTCOMES:
Anxiety at 12 hours | Evaluations will be made 12 hours after the intervention
  Anxiety will be evaluated by the Spanish version of the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). This scale has a score between 0 and 21 for either anxiety or depression with greater punctuation indicating a worse condition.
Anxiety at 48 hours | Evaluations will be made 48 hours after the intervention
  Anxiety will be evaluated by the Spanish version of the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). This scale has a score between 0 and 21 for either anxiety or depression with greater punctuation indicating a worse condition.
Anxiety at first visit | Evaluations will be made at first visit, between 10 and 12 days after the intervention.
  Anxiety will be evaluated by the Spanish version of the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). This scale has a score between 0 and 21 for either anxiety or depression with greater punctuation indicating a worse condition
Anxiety at one month | Evaluations will be made at one month after surgery.
  Anxiety will be evaluated by the Spanish version of the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). This scale has a score between 0 and 21 for either anxiety or depression with greater punctuation indicating a worse condition.
Postoperative nausea after surgery | At 12 hours after surgery
  The intensity of postoperative nausea will also be evaluated by the numerical rating scale (NRS)
Postoperative nausea at 24-48 hours | At 24-48 hours after surgery
  The intensity of postoperative nausea will also be evaluated by the numerical rating scale (NRS)
Post-operative complications | Up to one month.
  Post-operative complications such as seroma, infection and wound healing will be recorded.
Acupuncture adverse events | Up to one month.
  Adverse events possibly linked to acupuncture such as pain, hematomas etc. will be recorded.

IPD SHARING:
Plan to Share IPD: No